CLINICAL TRIAL: NCT02153047
Title: Multicentric Randomized Clinical Trial to Evaluate the Long-term Effectiveness of a Motivational Intervention Against Smoking, Based on the Information Obtained From Spirometry in Primary Care.
Acronym: RESET-ESPITAP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other); Catalan Institute of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI11/01962
Record Dates: First submitted 2014-05-28; First posted 2014-06-02 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-03

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Spirometry; Primary health care
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spirometry (Experimental): Will be given a brief but structured smoking cessation advice (according to the standards of the Tobacco Study Group of the Catalan Society of Family Medicine) together with a detailed and structured 20-minutes visit with details of the spirometry data (values of respiratory capacity and volumes referring on the theoretical)
  Interventions: Behavioral: Spirometry
- Brief smoking cessation advice (No Intervention): Will be given a brief but structured smoking cessation advice (according to the standards of the Tobacco Study Group of the Catalan Society of Family Medicine).

INTERVENTIONS:
Behavioral: Spirometry — Will be given a brief but structured smoking cessation advice (according to the standards of the Tobacco Study Group of the Catalan Society of Family Medicine) together with a detailed and structured 20-minutes visit with details of the spirometry data (values of respiratory capacity and volumes referring on the theoretical)
  Arms: Spirometry

SUMMARY:
There is controversy about the effectiveness of interventions based on spirometry for smoking cessation.

The investigators want to evaluate the effectiveness of motivational intervention performed by a doctor to obtain abstinence compared with normal practice in primary care.

This study, is the second half of what was began with ESPITAP study

DETAILED DESCRIPTION:
Design: Multicentric randomized clinical trial with two groups. Setting: 20 primary care centers inTarragona. Subjects: 1100 active smokers (consumption>10 packs/year) aged 35-70, seeking medical advice for any reason, with no exclusion criteria, will be randomized to receive the intervention or not.

Intervention: A 20-minutes visit with details of the spirometry data (values of respiratory capacity and volumes referring on the theoretical). The lung age index will be reported compared to chronological age to illustrate lung damage suffered as a result of tobacco consumption.

Measurements: Basal Spirometry. Structured questionnaire interviewed in the center at 0 and 12 months and telephone interview at 3 and 6 months. At 12 months, patients who stopped smoking will perform a CO test and if the CO exhaled will be <10ppm abstinence will be verified by determination of urinary cotinine.

Primary endpoint: Cessation of tobacco consumption at 12 months. Analysis: Data will be analyzed in the "intent to treat", the unit of analysis will be the smoker.

Expected Results: smoking cessation in the intervention group will exceed at least 5% the achieved by normal practice in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Active smokers (consumption>10 packs/year)

Exclusion Criteria:

* Active respiratory disease
* Practice of an espirometry on 12 months before
* Suffering of any chronic or terminal disorder
* Counterindication to undertake spirometry or that may hinder the performance of the spirometry test

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Cessation of tobacco consumption at 12 months. | 12 months

SECONDARY OUTCOMES:
Smoking reduction: self reported reduction | 12 Months
  Smoking reduction by self reported reduction

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Santigosa-Ayala, MD, Principal Investigator — Catalan Institute of Health; Francisco Martín-Luján, PhD, Study Director — Catalan Institute of Health; Rosa Sola-Alberich, MD, Study Chair — Catalan Institute of Health
Locations (1):
- Jordi Gol i Gurina Foundation, Barcelona, Spain

REFERENCES:
- [Derived] Martin-Lujan F, Santigosa-Ayala A, Palleja-Millan M, Rey-Renones C, Villalobos F, Sola R; researchers of the RESET study. Effectiveness of the spirometry-based motivational intervention to quit smoking: RESET randomised trial. Eur J Gen Pract. 2023 Dec;29(1):2276764. doi: 10.1080/13814788.2023.2276764. Epub 2023 Nov 7. PMID 37933978
- [Derived] Martin-Lujan F, Santigosa-Ayala A, Pinol-Moreso JL, Sorli-Aguilar M, Flores-Mateo G, Blade-Creixenti J, Basora-Gallisa J, Sola-Alberich R; RESET Study Group investigators. Multicentric randomized clinical trial to evaluate the long-term effectiveness of a motivational intervention against smoking, based on the information obtained from spirometry in primary care: the RESET study protocol. BMC Fam Pract. 2016 Feb 4;17:15. doi: 10.1186/s12875-016-0415-1. PMID 26846522